CLINICAL TRIAL: NCT07285499
Title: Prognostic Value of the CALLY Index in Intensive Care Patients Diagnosed With Sepsis: A Retrospective Cohort Study
Brief Title: Prognostic Value of the CALLY Index in Patients With Sepsis
Acronym: CALLY-SEP
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Oğuzhan Demirel, Resident Physician, Department of Anesthesiology and Reanimation, Ankara University
Other Study IDs: CALLY-Sepsis-2025-01
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Sepsis
Keywords: CALLY Index; Sepsis; Intensive Care Unit; Mortality; Acute Kidney Injury; SOFA Score; APACHE II
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis Cohort: Adult ICU patients diagnosed with sepsis according to Sepsis-3 criteria whose CALLY index values were obtained on day 0, day 3, and day 5.

SUMMARY:
This retrospective observational study evaluates the prognostic value of the C-reactive protein-albumin-lymphocyte (CALLY) index in adult patients with sepsis admitted to the intensive care unit (ICU). The CALLY index reflects inflammatory, nutritional, and immunologic status and may serve as a predictor of clinical outcomes.

CALLY Index values will be obtained on Day 0, Day 3, and Day 5 of ICU admission using routinely collected laboratory data. The primary objective is to determine the association between CALLY Index values and 30-day all-cause mortality. Secondary objectives include assessing the relationship between temporal CALLY changes and the development of acute kidney injury (AKI) within the first 7 days of ICU admission, as well as correlations between the Day-0 CALLY Index and established severity scores such as SOFA and APACHE II.

As this retrospective study uses existing electronic medical records, no additional procedures or interventions will be performed, and no added risk to patients is involved.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition characterized by a dysregulated host response to infection and is frequently associated with multiorgan dysfunction and high mortality. Early identification of patients at increased risk of poor outcomes remains a major challenge in critical care. The C-reactive protein-albumin-lymphocyte (CALLY) Index is a composite biomarker that reflects inflammatory, nutritional, and immune status. Although recent studies have explored the prognostic value of CALLY in critically ill populations, the significance of serial measurements and temporal changes in patients with sepsis has not been fully established.

This retrospective observational study will include adult patients diagnosed with sepsis according to Sepsis-3 criteria who were admitted to the intensive care unit (ICU) between January 2023 and December 2024. The CALLY Index will be calculated using the following formula:

Albumin (g/L) × lymphocyte count (10⁹/L) × 100 ÷ CRP (mg/L).

CALLY values will be obtained at predefined time points: Day 0 (within 2 hours of ICU admission), Day 3, and Day 5, extracted from the hospital's electronic medical record system.

The primary aim of the study is to evaluate the association between CALLY Index values and 30-day all-cause mortality. Secondary aims include assessing the relationship between temporal changes in CALLY (ΔCALLY₃-₀, ΔCALLY₅-₀, and linear trend slope) and the development of acute kidney injury (AKI) within the first 7 days of ICU admission, as well as examining correlations between the Day-0 CALLY Index and commonly used clinical severity scores, including SOFA and APACHE II.

All study data will be obtained retrospectively from the hospital's electronic records. No additional tests, procedures, or interventions will be performed. As the study utilizes existing clinical data without influencing patient management, it poses no additional risks to participants. The findings may support improved early risk stratification, monitoring of disease progression, and refinement of prognostic assessment in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Sepsis diagnosis meeting Sepsis-3 criteria
  * ICU stay ≥ 5 days
  * Complete CRP, albumin, and lymphocyte laboratory results available for days 0, 3, and 5

Exclusion Criteria:

* • Chronic Kidney Disease stage ≥3

  * Liver diseases including cirrhosis, chronic hepatitis, or hepatic failure
  * Hematologic diseases such as leukemia, lymphoma, MDS, or multiple myeloma
  * Rheumatologic diseases including SLE, rheumatoid arthritis, or systemic sclerosis
  * Use of immunosuppressive therapy
  * ICU stay shorter than 5 days
  * COVID-19 positive status
  * Missing laboratory data preventing calculation of CALLY index

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients diagnosed with sepsis and treated at Ankara University Medical Faculty Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
30-day All-Cause Mortality | 30 days after ICU admission
  Proportion of adult ICU patients with sepsis who die from any cause within 30 days after ICU admission.
  Vital status at 30 days will be obtained exclusively from the hospital electronic medical record system.
  Unit of measure: Percentage of participants. The CALLY Index will be calculated as: Albumin (g/L) × lymphocyte count (10⁹/L) × 100 ÷ CRP (mg/L).
  CALLY Index values measured on Day 0, Day 3, and Day 5 will be used as predictor variables in prognostic analyses, but they are not part of this outcome measure.

SECONDARY OUTCOMES:
Acute Kidney Injury (AKI) Development | Up to 7 days after ICU admission
  Occurrence of acute kidney injury (AKI) during ICU admission, defined according to KDIGO criteria (increase in serum creatinine or decrease in urine output). Unit of measure: Number of participants with AKI. CALLY Index values and temporal CALLY changes (ΔCALLY_3-0 and ΔCALLY_5-0) will be analyzed as predictor variables, but they are not part of this outcome measure.
Correlation Between CALLY Index Trends and Clinical Outcomes (Mortality and AKI) | Day 0 to Day 5 (first 5 ICU days)
  This outcome will assess the correlation between temporal changes in the CALLY Index and clinical outcomes (30-day mortality and AKI).
  CALLY Index will be calculated using the formula:
  Albumin (g/L) × lymphocyte count (10⁹/L) × 100 ÷ CRP (mg/L).
  Temporal CALLY changes will include:
  * ΔCALLY₃-₀ (difference between Day-3 and Day-0 values),
  * ΔCALLY₅-₀ (difference between Day-5 and Day-0 values),
  * CALLY trend slope (calculated using linear regression across Day-0, Day-3, and Day-5 values).
  These variables will be used as predictor variables in prognostic analyses. Unit of measure: Correlation coefficient
Correlation Between Day-0 CALLY Index and Severity Scores (SOFA, APACHE II) | Day 0 (within 2 hours of ICU admission)
  This outcome will assess the correlation coefficient between the Day-0 CALLY Index and severity scores (SOFA and APACHE II).
  The CALLY Index will be calculated as: Albumin (g/L) × lymphocyte count (10⁹/L) × 100 ÷ CRP (mg/L), using laboratory results obtained within 2 hours of ICU admission (Day 0).
  SOFA score will be measured using the standard Sequential Organ Failure Assessment scale (range: 0-24).
  APACHE II score will be calculated using the established APACHE II scoring system (range: 0-71).
  Unit of measure: Correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine - Intensive Care Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No